CLINICAL TRIAL: NCT00958321
Title: Prospective Evaluation of PET-CT Scan in Patients With Non-operable or Non-resectable NSCLC Treated by Radical 3-Dimensional Conformal Radiation Therapy
Brief Title: Positron Emission Tomography and Computed Tomography in Planning Treatment for Patients Undergoing 3-Dimensional Conformal Radiation Therapy for Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery. ICORG 06-35
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low levels of recruitment
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTRIAL-IE (ICORG)06-35; CTRIAL-IE (ICORG) 06-35; EU-20925
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer; malignant pleural effusion; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Adenocarcinoma of Lung; Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Fluorodeoxyglucose F18

ARMS (1):
- 3-DCRT (Experimental): Patients will receive a total dose of 60-66 Gy in 30-33 fractions with 3-DCRT
  Interventions: Procedure: computed tomography; Radiation: 3-dimensional conformal radiation therapy; Radiation: fludeoxyglucose F 18; Radiation: radiation therapy treatment planning/simulation

INTERVENTIONS:
Procedure: computed tomography
Radiation: 3-dimensional conformal radiation therapy
Radiation: fludeoxyglucose F 18
Radiation: radiation therapy treatment planning/simulation

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography and computed tomography, may help learn the extent of disease and allow doctors to plan 3-dimensional conformal radiation therapy.

PURPOSE: This phase II trial is studying the side effects of positron emission tomography and computed tomography and to see how well it works in planning treatment for patients undergoing 3-dimensional conformal radiation therapy for non-small cell lung cancer that cannot be removed by surgery.

This is a clinical study, as the patient will be treated using the PET-CT-GTV: - The pilot study is investigating the technological feasibility - The Phase II study will be a 2-stage Phase II study

DETAILED DESCRIPTION:
Pilot Study- Primary Objectives:

* Prospective evaluation of the technical feasibility of integrating PET-CT fusion in St Luke's Hospital
* Rate of PET-CT Scan based treatment delivery

Pilot Study- Secondary Objectives:

-Comparison of GTV, PTV and OAR DVHs between conventional 3-DCRT plan and PET-CT based 3-DCRT plan.

Phase II Study- Primary Objective:

-The safety of PET-CT scan based radiotherapy, with regard to loco-regional disease control.

Phase II Study- Secondary Objectives:

-Comparison of GTV, PTV and OAR DVHs between conventional 3-DCRT plan and PET-CT based 3-DCRT plan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven (biopsy or cytology) NSCLC (SCC, Adenocarcinoma, Large Cell)
* TNM clinical non-operable stage I/II and non-resectable stage IIIa/b without pleural effusion
* Measurable disease
* No other malignancy, except non-melanomatous skin cancer, within 5 years prior to participation in this study; the disease-free interval from any prior carcinoma must be continuous
* Patient suitable for radical 3-DCRT
* ECOG-Performance status ≤ 2 / KPS > or equal to 60
* Weight loss <10% within the 3 months prior to diagnosis
* No prior radiotherapy to the thorax
* Patient is suitable for lung-board immobilisation
* No chemotherapy received prior to planning PET-CT scan
* Age 18 and over
* Provision of written informed consent

Exclusion Criteria:

* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial or if it is felt by the research / medical team that the patient may not be able to comply with the protocol.
* FEV1 < 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-03; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Rate of successful delivery of PET-CT scan based 3-D conformal radiotherapy (Pilot) | 2016
Rate of loco-regional recurrence outside the PET-CT planning target volume (PTV) but within conventional 3-D PTV (Phase II) | 2016

SECONDARY OUTCOMES:
Acute and long-term radiation-induced toxicity | 2016
Comparison of dose delivery to organs at risk, according to planning method | 2016

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, MD, Principal Investigator — Saint Luke's Hospital
Locations (1):
- St Luke's Radiation Oncology Network, Dublin, Ireland